CLINICAL TRIAL: NCT03619330
Title: Effects of Liraglutide and Testosterone Replacement Therapy on Features of Hypogonadism and Weight Loss in Obese Men With Persistent Features of Hypogonadism.
Brief Title: Testosterone Replacement Therapy and Liraglutide Effects on Weight Loss in Hypogonadism.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, professor, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TESTOSTERON
Record Dates: First submitted 2018-07-16; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Hypogonadism; Obesity
MeSH Terms: conditions — Hypogonadism; Obesity | interventions — Liraglutide; Solutions; Injections; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- liraglutide (Active Comparator): In the LIRA group liraglutide was initiated at a dose of 1.2 mg injected sc once per day and increased to 3 mg/day after 1 week.
  Interventions: Drug: liraglutide
- testosterone (Active Comparator): In the ANDRO group testosterone was initiated at a dose of 50 mg in a gel form once daily.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: liraglutide — In the liraglutide group liraglutide was initiated at a dose of 1.2 mg injected sc once per day and increased to 3 mg/day after 1 week.
  Other Names: Victoza 6 mg/ml solution for injection in pre-filled pen
  Arms: liraglutide
Drug: Testosterone — In the testosterone group Androtop gel 5 grams (50 mg of testosterone) was applied once a day on a dry skin.
  Other Names: Androtop gel
  Arms: testosterone

SUMMARY:
The purpose of this study was to compare the effects of liraglutide and testosterone replacement therapy on features of hypogonadism and weight loss in obese men with persistent features of hypogonadism after unsuccessful lifestyle measures.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The main outcome was improvements of symptoms related to hypogonadism | Patients were screened and asked for symptoms at the beginning and every 4 weeks for 16 weeks of the study.
The main outcome was change testosterone level. | Patient's blood was drawn at the base point and every four weeks during 16 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Concentrations of testosterone was measured in nmol/L.
the main outcome was change in gonadotropin levels. | Patient's blood was drawn at the base point and every four weeks during 16 weeks of clinical trial.

SECONDARY OUTCOMES:
The secondary outcome was change in body weight. | Patient's body weight in kilograms were measured at the base point and every four weeks during the 16 weeks of clinical trial.
The secondary outcome was change in waist circumference. | Patient's waist circumference was measured at the basepoint and every four weeks during 16 weeks of clinical trial.
  Patient's waist circumference was measured in centimeters.

OTHER OUTCOMES:
The other outcomes was changes changes in fasting concentrations of glucose. | Patient's fasting blood was drawn at the basepoint and and the end of the 16 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Concentrations of fasting glucose was measured in mmol/L.
Other outcome was change in fasting concentration of insulin. | Patient's fasting blood was drawn at the basepoint and and the end of the 16 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Fasting concentrations of insulin was measured in mU/L.
Other outcome was change in HOMA IR index for insulin resistance. | Patient's fasting blood was drawn at the basepoint and and the end of the 16 weeks of clinical trial.
  HOMA IR index was calculated as fasting plasma glucose times fasting plasma insulin devided by 22.5

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janez, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia